CLINICAL TRIAL: NCT04635709
Title: Effect of Behavioral Therapy Versus Interferential Current on Bladder Dysfunction in Patients With Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, walaa M Ragab, DR, Taibah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: taibahu
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Bladder Dysfunction on Patients With Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behavioral therapy (Experimental): applying biofeedback training on the pelvic floor muscles
  Interventions: Device: biofeedback training and interferential therapy
- interferential therapy (IF) (Experimental): Interferential current was applied to the body using four surface electrodes placed on the lower abdomen and lower buttocks.
  Interventions: Device: biofeedback training and interferential therapy

INTERVENTIONS:
Device: biofeedback training and interferential therapy — compare the effect of applying both types of devices on the pelvic floor muscles

SUMMARY:
study the effect of behavioral therapy and interferential current on management of bladder dysfunction in patients with multiple sclerosis

DETAILED DESCRIPTION:
Fifty patients with multiple sclerosis (MS) (secondary progressive type SPMS) suffering from bladder dysfunction were divided equally into two groups randomly; Group A received biofeedback training (behavioral therapy) while group B received interferential training. Both groups were assessed by urodynamics for detrusor pressure and maximum flow rate before and after eight weeks of behavioral therapy and interferential training.

Data analysis was managed using SPSS for windows, version 22 (SPSS, Inc., Chicago, IL). The current test involved two independent variables. The first one was the (tested group); between subject factors which had two levels (group A received behavioral therapy and group B who received IF ) .The second one was the (measuring periods); within subject factor which had two levels (pre, post). In addition, this test involved two tested dependent variables (detrusor pressure and maximum flow rate ) .T independent and dependent tests were used to compare between and within groups respectively. Data was considered statistically significant when P < .05

ELIGIBILITY:
Inclusion Criteria:

* All the patients were referred by a neurologist and the diagnosis was confirmed by the Magnetic Resonance Image (MRI).The duration of being diagnosed as SPMS for both groups were between one to two years. All the selected patients had normal mental examination according to mini mental scale .Also, all the selected patients were medically stable.

Exclusion Criteria:

* Patients with any other neurological deficits or orthopedics abnormalities or with auditory dysfunction were excluded from this study. Patients with history of bladder dysfunctions before the diagnosis of MS or attaining any attack during the treatment period were also excluded.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male patients with multiple sclerosis complaining of bladder dysfunctions
Enrollment: 50 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Detruser pressure between and within groups | eight weeks
  test it by urodynamic test before and after management
Maximum flow rate between and within groups | eight weeks
  test it by urodynamic test before and after management

CONTACTS AND LOCATIONS:
Overall Officials: walaa M Ragab, PHD, Principal Investigator — Taibah University ,saidi arab
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF